CLINICAL TRIAL: NCT03690739
Title: Trabectedin/PLD Versus Continuation of Platinum-based Chemo-therapy in Patients With Disease Stabilization and no Symptom Benefit Under Platinum-based Chemotherapy for Recurrent Ovarian Cancer
Brief Title: Evaluation of Symptom Benefit Rate of Trabectedin/PLD in Patients With Recurrent Ovarian Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient Recruitment
Sponsor: AGO Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AGO-OVAR 2.32
Record Dates: First submitted 2018-09-26; First posted 2018-10-01 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Recurrent Ovarian Carcinoma
Keywords: Symptom Benefit
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Gemcitabine; Bevacizumab; 1-dodecylpyridoxal; Paclitaxel; Trabectedin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platinum-based chemotherapy (Active Comparator): According to the investigator's discretion
  Interventions: Drug: Carboplatin; Drug: Gemcitabine; Drug: Bevacizumab; Drug: PLD; Drug: Paclitaxel; Drug: Cisplatin
- PLD + Trabectedin (Active Comparator): PLD 30 mg/m² + Trabectedin 1.1 mg/m² q21
  Interventions: Drug: PLD; Drug: Trabectedin

INTERVENTIONS:
Drug: Carboplatin — Administration according to investigator's discretion
  Arms: platinum-based chemotherapy
Drug: Gemcitabine — Administration according to investigator's discretion
  Arms: platinum-based chemotherapy
Drug: Bevacizumab — Administration according to investigator's discretion
  Arms: platinum-based chemotherapy
Drug: PLD — Administration according to investigator's discretion
  Arms: platinum-based chemotherapy
Drug: Paclitaxel — Administration according to investigator's discretion
  Arms: platinum-based chemotherapy
Drug: PLD — Administration 30 mg/m² q21
  Arms: PLD + Trabectedin
Drug: Trabectedin — Administration 1.1 mg/m² q21
  Arms: PLD + Trabectedin
Drug: Cisplatin — Administration according to investigator's discretion
  Arms: platinum-based chemotherapy

SUMMARY:
This is an open-label, prospective, randomized, controlled, parallel group, multi-center phase III trial to evaluate the Symptom Benefit Rate of trabectedin/PLD in patients with recurrent ovarian cancer who achieve a stabilization of disease after 3 cycles of platinum-based reinduction therapy and with no clinical benefit.

DETAILED DESCRIPTION:
Approximately 330 patients will be randomized in a 1:1 ration to the treatments specified below:

Arm A - Platinum-based chemotherapy according to investigator's discretion Arm B - Pegylated liposomal doxorubicin 30 mg/m² + Trabectedin 1.1 mg/m² (q3w)

ELIGIBILITY:
Inclusion Criteria:

1. Females aged ≥ 18 years at time of signing informed consent form.
2. Histologically proven diagnosis of cancer of the ovary, the fallopian tube or primary peritoneal cancer.
3. Measurable or non-measurable disease (according RECIST v1.1) or CA-125 assessable disease (according GCIG criteria) or histologically proven diagnosis of relapse.
4. Platinum-treatment free interval (TFIp) > 6 months prior to cycle 1 day 1 of reinduction therapy.
5. Disease stabilization without remission or progression ac-cording to RECIST or GCIG criteria after three cycles of platinum-based chemotherapy for recurrent disease.
6. Symptomatic disease at time of baseline abdominal/GI symptom scale score >15 (EORTC QLQ-OV28)
7. Completion of EORTC QLQ-OV28 at Baseline within 7 days prior to treatment start.
8. Patients should have received previously a taxane derivative.
9. ECOG performance status ≤ 2.
10. Life expectancy of at least 12 weeks.
11. Adequate bone marrow, renal and hepatic function defined as:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
    * Platelet count ≥ 100 x 10^9/L
    * Hemoglobin ≥ 9.0 g/dL
    * Serum creatinine ≤1.5 mg/dL (≤ 132.6 µmol/L) or creatinine clearance ≥ 60 mL/min
    * Creatine phosphokinase (CPK) ≤ 2.5 x ULN
    * Serum aspartate aminotransferase (AST, SGOT) or alanine aminotransferase (ALT, SGPT) ≤ 2.5 x ULN (≤ 5 x ULN in the presence of liver metastases)
    * Alkaline phosphatase (ALP) ≤ 2.5 ULN
    * Serum bilirubin ≤ ULN
    * Albumin ≥ 25 g/l
12. Participation in an informed consent discussion with the appropriate trial-related health care representative, full understanding of the implications and constraints of the protocol, and provision of written informed consent prior to the commencement of the trial-related procedures.
13. Geographically accessibility for treatment and follow-up.
14. For women of childbearing potential (WOCBP): agreement to remain abstinent (refrain from heterosexual inter-course) or use a contraceptive method with a failure rate of < 1 per-centage per year during the treatment period and for at least six months after administration of the last dose of chemo-therapy. A woman is considered to be of childbearing po-tential if she is postmenarcheal, has not reached a post-menopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries, fal-lopian tubes, and/or uterus). Examples of contraceptive methods with a failure rate of < 1 percentage per year in-clude but are not limited to bilateral tubal ligation and/or oc-clusion, male sterilization, and intrauterine devices, and nor-mal and low dose combined oral pill plus male condom or Cerazette (desogestrel) plus male condom. Cerazette is currently the only highly efficacious progesterone based pill. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation meth-ods) and withdrawal are not acceptable methods of contra-ception.

Exclusion Criteria:

1. Ovarian tumors of low malignant potential (e.g. borderline tumors).
2. Non-epithelial ovarian or mixed epithelial/non epithelial tumors (e.g. mixed Müllerian tumors).
3. Patients with an objective response in terms of a partial or complete remission or alternatively progressive disease ac-cording to RECIST or GCIG criteria after three cycles of platinum-based reinduction chemotherapy.
4. Patients who have received previous radiotherapy for ovarian cancer.
5. History of congestive heart failure (NYHA classification > 2, even if medically con-trolled).
6. History of myocardial infarction within the last six months (documented or by electrocardiogram).
7. History of atrial or ventricular arrhythmias.
8. Impaired liver function, hyperbilirubinemia, Serum creatinine >1.5 mg/dL or > 132.6 μmol/L or creatinine clearance < 60 mL/min, left ventricular ejection fraction < 45 %.
9. Severe active or uncontrolled infection.
10. Concurrent severe medical problems unrelated to malignancy, which would significantly limit full compliance with the trial or expose the patient to extreme risk or decreased life expectancy.
11. Patients with known hypersensitivity to the active substance or their compounds related to trabectedin or PLD and patients with known hypersensitivity to one of active substances or one of their compounds used in platinum-based chemotherapy as described in the Summaries of Medicinal Products.
12. Patients with potential risks according to contraindication, warnings or interactions of the used chemotherapeutic agents as stated in the SmPCs are not eligible for participation in this trial.
13. Patients with contraindication regarding CT or MRI (only in case of contrast allergy) are excluded.
14. Women of childbearing potential (WOCBP) not using highly effective contraceptive methods.
15. Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Symptom Benefit Rate | from Baseline to 8 or 9 weeks after randomization, assessed at each visit
  Proportion of patients achieving a symptom benefit defined as an at least 10-point improvement according to EORTC QLQ-OV28; EORTC QLQ-OV28 is a questionnaire regarding Quality of Life specialized for Ovarian Cancer with points from 1 till 4 for each of the 28 questions (1=not at all, 2=a little, 3=quite a bit, 4=very much). Points will be summarized.

SECONDARY OUTCOMES:
Time until definitive deterioration (TUDD ) | from Baseline until 24 months after randomization, assessed up to 54 months at each visit
  TUDD is defined as time from baseline until the first decrease in EORTC QLQ-C30 score ≥ 10 points (or 20 points) as compared at baseline; EORTC QLQ-C30 is a questionnaire regarding Quality of Life specialized for Cancer with points for each of the 30 questions (1=not at all, 2=a little, 3=quite a bit, 4=very much). Points will be summarized.
Progression-free survival (PFS) | PFS is defined as time from randomization to disease progression according to RECIST v1.1, to death from any cause or to start of a new treatment (whichever occurs first), assessed up to 54 months
  Progressive disease is based on investigator assessment using RECIST v1.1
Progression-free survival (PFS) rate at 6 months | PFS is defined as time from randomization to disease progression according to RECIST v1.1, to death from any cause or to start of a new treatment (whichever occurs first) after six months
  Progressive disease is based on investigator assessment using RECIST v1.1
Response Rate (RR) | from randomization until patients achieving complete response (CR) or partial response (PR) as best overall response, assessed up to 54 months
  RR is based on investigator assessment using RECIST v1.1
Global Health Status | from baseline to end of treatment, assessed up to 54 months at each visit
  based on Quality of Life; EORTC QLQ-C30 and EORTC QLQ-OV 28 are questionnaires for Quality of Life with points for each of the 30 or 28 questions (1=not at all, 2=a little, 3=quite a bit, 4=very much). Points will be summarized.
Overall Survival (OS) | OS is defined as the time from randomization to death from any cause, assessed up to 54 months
  regular patient contact during the trila regarding life status

CONTACTS AND LOCATIONS:
Overall Officials: Felix Hilpert, MD, PhD, Study Chair — Mammazentrum am Krankenhaus Jerusalem, Hamburg
Locations (29):
- Germany (29):
  - Klinikum Aschaffenburg-Alzenau, Aschaffenburg, Bavaria
  - Hochtaunus-Kliniken, Bad Homburg
  - Sozialstiftung Bamberg, Bamberg
  - Evangelisches Krankenhaus Bergisch Gladbach, Bergisch Gladbach
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsfrauenklinik Bonn, Bonn
  - Schwerpunktpraxis für Onkologie / Hämatologie, Bottrop
  - Frauenärzte Casparistraße, Braunschweig
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Evang. Kliniken Essen-Mitte, Essen
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Universitätsmedizin Greifswald, Greifswald
  - Mammazentrum Hamburg am Krankenhaus Jerusalem, Hamburg
  - Klinikum Itzehoe, Itzehoe
  - ViDia Christliche Kliniken Karlsruhe, Karlsruhe
  - Klinikum Ludwigsburg, Ludwigsburg
  - Klinikum Magdeburg, Magdeburg
  - Katholisches Klinikum Mainz, Mainz
  - Universitätsfrauenklinik Mannheim, Mannheim
  - Klinikum Memmingen, Memmingen
  - Klinikum rechts der Isar, München
  - Kliniken des Landkreises Neumarkt, Neumarkt
  - Universitätsklinik für Innere Medizin, Onkologie und Hämatologie, Oldenburg
  - Klinikum Ernst von Bergmann, Potsdam
  - Agaplesion Diakonieklinikum Rotenburg, Rotenburg (Wümme)
  - Thüringen Kliniken "Georgius Agricola", Saalfeld
  - g.Sund Gyn. Kompetenzzentrum, Stralsund
  - Kreiskrankenhaus "Johann Kentmann", Torgau
  - Helios Dr. Horst Schmidt Kliniken, Wiesbaden